CLINICAL TRIAL: NCT06399549
Title: Effects of Dead Bug vs. Mc Gill Exercises on Pain, Quality of Life and Core Stability in Patient With Chronic Nonspecific Low Back Pain
Brief Title: Effects of Dead Bug vs. Mc Gill Exercises on Pain, QOL and Core Stability in Patient With Chronic Nonspecific LBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall19/561
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dead bug exercise (Experimental)
  Interventions: Diagnostic Test: Dead bug exercise
- The McGill Curl Up (Experimental)
  Interventions: Diagnostic Test: The McGill Curl Up

INTERVENTIONS:
Diagnostic Test: Dead bug exercise — the participant in supine, lying on a mat with shoulders, hip joints and knees flexed to 90°. With the lumbopelvic region being maintained in the neutral position, the participant will be instructed to draw in the abdomen, lower two contra lateral limbs (opposite arm and leg) toward the floor, hold for the stipulated time, then return to starting position. The same movement will be repeated with the opposite limbs. In the DBG, both pairs of limbs will be moved an equal number of times withinthe stipulated time. The patients in both groups will perform the corresponding exercises 3 days a week for a period of 3 weeks and a rest interval of 2 minutes between exercises along with conventional physiotherapy exercises.
  Arms: Dead bug exercise
Diagnostic Test: The McGill Curl Up — Lie down on your back. Extend one leg and bend the knee of the other leg. The Side Bridge. Lie on your side, with your forearm on the floor and elbow underneath your shoulder.
  The Bird Dog. Assume a hands-and-knees position on the floor. The patients in both groups will perform the corresponding exercises 3 days a week for a period of 3 weeks and a rest interval of 2 minutes between exercises along with conventional physiotherapy exercises. The exercise program includes a warm-up session of five exercises (awareness of the back, pelvic tilt, lumbar rotation, arm movements, whole-body movement in standing), well-known exercises targeting the muscles of the back extensors, abdominals, lateral buttocks, trunk rotators, posterior buttocks, leg muscles, oblique abdominals (e.g. the plank, diagonal arm and leg lift), as well as exercises for flexibility. The exercises will be taught to the patients at the end of the first session in both groups.
  Arms: The McGill Curl Up

SUMMARY:
Low back pain is one of the most common conditions for which patients are sent to physiotherapy clinics. 84% of people have experienced it at least once in their lifetime, and over 50% have experienced it more than once, according to research. However, diagnosis and, in particular, the provision of specialized back pain therapy remain difficult.

DETAILED DESCRIPTION:
This study aims to compare the effects of dead bug vs. Mc Gill exercises on pain, quality of life and core stability in patient with chronic nonspecific low back pain. It will be a randomized clinical trial study. The sample size of study will be 44 participants (22 in each group). Data will be collected from Azra Naheed Hospital. Data will be collected within 6 months after approval of synopsis. Group A will follow dead bug exercises and Group B will follow Mc Gill exercises (Curl up, Side Bridge and Bird Dog). The patients in both groups will be performed the corresponding exercises 3 days a week and 10 repetitions of each exercise for a period of 6 weeks and a rest interval of 2 minutes between exercises. The exercises will be taught to the patients at the end of the first session in both groups. The data will be analyzed using SPSS version 24 for Windows software. Statistical significance will be set at P ≤ 0.05. Normality of data will be assessed through Kolmogorov-smirnov test. Difference between pre-treatment and post-treatment readings will be calculated using Paired sample t-test for parametric data. For non-parametric data Wilcoxon test will be used. Independent sample t test will be used for parametric data and Mann Whitney test will be used for non parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50 years
* Patient with the history of 3 months nonspecific low back pain
* Pain intensity (3-7) according to VAS score

Exclusion Criteria:

* Spinal stenosis
* Neurological dysfunction
* Systemic disease
* Pregnancy
* Infections
* Carcinoma
* Any fracture or deformity

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-09 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
VA | 6 Months
  Visual Analogue Scale (VAS) is one of the pain rating scales 10 for worse and 0 for no pain

SECONDARY OUTCOMES:
SF36 | 6 Months
  The Short Form 36 Health Survey (SF-36) is a commonly used scale to assess HRQoL. Thirty-six questions divided into 8 dimensions. Higher scores are associated with better HRQOL. The SF-36 health-related quality of life questionnaire is well applied to assess the quality of life due to its reliability or validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Ganga Ram Hospital Physiotherapy department , Mozang, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No